CLINICAL TRIAL: NCT02881619
Title: Preemptive Use of Etodolac on Tooth Sensitivity Caused by In-office Bleaching: a Randomized, Triple-blind, Controlled Clinical Trial
Brief Title: Etodolac and Post-bleaching Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flavia Pardo Salata Nahsan (Other)
Responsible Party: Sponsor-Investigator, Flavia Pardo Salata Nahsan, Clinical Professor, Universidade Federal de Sergipe
Organization: Universidade Federal de Sergipe (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UFS
Record Dates: First submitted 2016-08-04; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Medicaments Substances in Therapeutic Use
Keywords: Tooth bleaching
MeSH Terms: interventions — Etodolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo - (inert content)
  Interventions: Drug: Placebo
- Experimental - (Experimental): 400 mg of NAISE etodolac
  Interventions: Drug: Etodolac

INTERVENTIONS:
Drug: Etodolac — The patient will receive a single-dose of Etodolac (400 mg) one hour before the bleaching procedure.
  Arms: Experimental -
Drug: Placebo — The patient will receive a single-dose of placebo one hour before the bleaching procedure.
  Arms: Placebo

SUMMARY:
Objectives: This study will determine the effectiveness of preemptive administration of etodolac on risk and intensity of tooth sensitivity caused by in-office bleaching using 35% hydrogen peroxide.

Materials and Methods: Fifty patients will be selected for this triple-blind, randomized, cross-over, placebo-controlled clinical trial. Etodolac (400 mg) or placebo will be administrated in a single-dose 1 hour prior to bleaching procedure. The whitening treatment with 35% hydrogen peroxide will be carried out in two sessions with a 7-day interval. Tooth sensitivity will be assessed before, during and 24 hours after the procedure using analog visual and verbal scales. Color alteration will be assessed by a bleach guide scale 7 days after each session. Relative risk to sensitivity will be calculated and adjusted by session; while comparison of overall risk will performed by McNemar's test. Data on the sensitivity level for both scales and color shade will be subjected to the Friedman, Wilcoxon and Mann-Whitney tests, respectively (α = 0.05).

DETAILED DESCRIPTION:
Methods & Materials:

This clinical trial was approved by the Scientific Review Committee and by the Committee for the Protection of Human Subjects of the local university (CAAE 37578714.4.0000.5546).

Trial design:

This study will be a randomized, triple-blind, placebo-controlled clinical trial with a cross-over design. The patients included will be submitted to two in-office bleaching sessions receiving placebo (control) or etodolac prior to the bleaching procedure; while different treatments will be allocated for each session. A delay of 1 week between the sessions (wash-out) will be established. The study will be conducted at the clinic of the School of Dentistry of the local university from November 2014 to July 2015.

Participants:

Patients included in this clinical trial will be at least 18 years old with good oral health. Patients with any of the six upper anterior teeth with caries, restoration, severe discoloration (e.g., stains caused by tetracycline), enamel hypoplasia, gingival recession, dentin exposure, pulpitis, or endodontics will be excluded. Participants submitted to previous bleaching procedures, presenting prior tooth sensitivity, known allergy to any component of medication used in the study, pregnant or breastfeeding will be also excluded. Only patients presenting all six upper anterior teeth with shade mismatching with 2.5 M2 (Vita Bleachguide 3D-Master scale, Vita-Zahnfabrik, Bad Sackingen, Germany) or darker will be included.

Sample Size Calculation:

The sample calculation will be based on the primary binary outcome (sensitivity risk 24 hours after the procedure) for superiority trial. Power of the test will be set at 80%, considering a type I error of 0.05; risk to tooth sensitivity of 90%, based on a prior study using similar bleaching agent, while a reduction around 30% with the treatment will be expected. The calculation resulted in fifty patients.

Randomization:

A randomized list will be computer-generated by a person not involved in intervention or evaluation. The participants were defined as blocks in the randomization process, where the sequence of treatment (placebo or etodolac) will be randomly set for each block by using computer-generated tables (www.sealedenvelope.com). The sequence will be inserted into sealed envelopes numbered from 1 to 50 that were opened by the operator only at the moment of the intervention. The patients were numbered according to the sequence of enrollment. Neither the participant nor the operator knew the group allocation determining blinding to the protocol.

Baseline evaluation:

Prior to bleaching procedure, the teeth will be cleaned using rubber cups associated to pumice and water. The shades of six upper anterior teeth will be assessed on a baseline using the bleach guide scale. The color analysis will be carried out by two previously calibrated evaluators. The two evaluators presented superior color matching competency according to the ISO (International Organization for Standardization) 28642:2011. The shades' tabs selected will be converted to scores ranging from 1 (whiter shade - 0M1) to 15 (darker shade - 5M3).

Considering a possible effect of dental anxiety on sensitivity reported by patients, the Corah's Dental Anxiety Scale will be used to determine the level of anxiety of each patient related to the procedure [26]. Each answer to the survey instrument will be scored on a scale from 1 to 5 (four questions); and the sum of scores will be used to determine the level of anxiety: low will be lower than 12, moderate will be between 12 and 14, and high will be higher than 14.

Intervention:

One-hour prior to each bleaching session, the patients will receive a capsule containing 400 mg of NAISE etodolac or 400mg of placebo (inert content), according to the randomization, while the capsules will present the same appearance. The capsules with similar presentation will be manufactured by a person not involved in intervention or evaluation and will be placed into two bottles identified by letters according to treatment. Neither the operators responsible for intervention and evaluation nor the patients knew the content of each capsule.

A light-cured resin dam will be applied (Top Dam, FGM, Joinville, SC, Brazil) on the gingival tissue corresponding to the teeth to be bleached. A 35% hydrogen peroxide based bleaching agent (Whiteness HP Blue, FGM, Joinville, SC, Brazil) will be mixed and applied on the vestibular surface of teeth, remaining for 40 minutes. After this time, the bleaching agent will be removed. A second session will beas carried out after 1 week following the same procedures. At this time, the patient received a single-dose capsule containing etodolac or placebo (different from the ones received at first session) 1 hour before the procedure.

Evaluations:

The tooth sensitivity reported by patients will be assessed using a visual analog scale (VAS) and verbal rating scale (VRS). The VAS consisted of a scale 10 cm in length ranging from green (absence of pain) to red (unsupportable pain). The patient set his or her level of sensitivity by pointing to the color corresponding to this level, while the distance from this point to the green border will be recorded. For VRS, the patient reported his or her level of sensitivity based on scores: 0 = none, 1 = light, 2 = moderate, 3 = considerable and 4 = severe. The tooth sensitivity will be assessed during the bleaching, immediately after bleaching agent removal and after 24 hours. For this last assessment, only the VRS will be used. One week after each session the tooth color will be evaluated again using the same procedure described previously.

Statistical Analysis:

The demographic data from patients will be analyzed to determine age, gender, and anxiety level for each allocation sequence. Comparisons between the allocation sequences will be performed by the Mann-Whitney test (age) and Fisher's exact (gender) and chi-square (anxiety level) tests.

Based on presence of any tooth sensitivity (scores different from 0 for VRS), the absolute risk, odds ratio and relative risk will be calculated regarding the treatments for each moment of evaluation/session of bleaching, as well as its confidence intervals (95%). For each moment, differences on presence/absence ratios will be analyzed by Fisher's exact test. For the overall risk related to each treatment, the odds ratio will be adjusted to independent variable "session of bleaching" using the Mantel-Haenszel statistic. The homogeneity of odds ratios will be analyzed by the Breslow-Day and Tarone's tests. Following, the odds ratio estimated will be converted to relative risk and the overall presence/absence ratios will be analyzed by the McNemar's test, considering the study design (cross-over).

For VRS, the data from scores observed in each time of evaluation/session of bleaching will be submitted to the Mann-Whitney rank sum test. Despite the measurement of tooth sensitivity using VAS giving a continuous outcome, data assessed with this scale did not show a normal distribution (Shapiro-Wilk's test). Thus, data from VAS will be also analyzed by the Mann-Whitney rank sum test, while one test per time of evaluation will be carried out.

For color evaluation, comparisons between the sequences of treatment will be performed using the Mann-Whitney rank sum test. The Friedman test followed by Dunn's post hoc test will be used to analyze the difference between the moments of evaluation for each sequence of treatment. All statistical analyses will be performed adjusting the initial significance level (α = 0.05) by Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this clinical trial will be at least 18 years old with good oral health. . Only patients presenting all six upper anterior teeth with shade mismatching with 2.5 M2 (Vita Bleachguide 3D-Master scale, Vita-Zahnfabrik, Bad Sackingen, Germany) or darker will be included.

Exclusion Criteria:

* Patients with any of the six upper anterior teeth with caries, restoration, severe discoloration (e.g., stains caused by tetracycline), enamel hypoplasia, gingival recession, dentin exposure, pulpitis, or endodontics will be excluded. Participants submitted to previous bleaching procedures, presenting prior tooth sensitivity, known allergy to any component of medication used in the study, pregnant or breastfeeding will be also excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Risk to the tooth sensitivity | During the bleaching treatment.
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Level of tooth sensitivity - during procedure | During the Bleaching procedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe.
Risk after tooth sensitivity - after the procedure | 24 hours after the Bleaching procedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated
Level of tooth sensitivity - after the procedure | 24 hours after the Bleaching procedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Pardo Salata Nahsan, Principal Investigator — Universidade Federal de Sergipe

IPD SHARING:
Plan to Share IPD: No